CLINICAL TRIAL: NCT05694208
Title: The Effect of Mobile-Based Education Given to Patients Undergoing Gynecological Oncology Surgery on Quality of Life
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Çisem Baştarcan, PhD student, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CBastarcan
Record Dates: First submitted 2023-01-12; First posted 2023-01-23 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Gynecologic Cancer
Keywords: Gynecological oncology; Mobile application; Nursing care

STUDY DESIGN:
Intervention Model Description: The women included in the study sample will be divided into two groups as experimental and control groups according to randomization. Experimental group; the group to be trained. control group; This is the group in which no attempt will be made other than data collection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The patients in the experimental group will use the mobile-based care support application developed within the scope of the research.
  Interventions: Behavioral: Education Group
- Control Group (No Intervention): It is the group in which no intervention will be made other than data collection.

INTERVENTIONS:
Behavioral: Education Group — In the first pre-operative interview at the gynecological oncology outpatient clinic of the relevant hospital, the purpose of the research will be explained to the patients and an informed consent form will be filled. The patients in the experimental group will use the mobile-based care support application developed within the scope of the research.
  Arms: Experimental group

SUMMARY:
This study was planned in a randomized controlled prospective experimental design in order to determine the effect of mobile-based education given to patients undergoing gynecological oncology surgery on quality of life.

Research Hypotheses:

H1. Education given with mobile application in gynecological oncology patients positively affects symptom control of patients.

H2. The education given with the mobile application in gynecological oncology patients positively affects the quality of life of the patients.

DETAILED DESCRIPTION:
Power analysis was conducted to determine the number of people to be included in the study. The power of the test was calculated with the G*Power 3.1 program. As a result of the power analysis, the sample size should be 50, 25 experimental and 25 control groups, at 95% power, 5% significance level, and 0.690 effect size (df=24; t=1,710). In the research, it was aimed to reach a total of 70 women, 35 people in each group, considering the high power of the test and the losses.

Introductory Information Form, Symptom Evaluation Form, Functional Assessment of Cancer Therapy-General (FACT-G) and Turkish-Computer System Usability Questionnaire (T-CSUQ- SV) planned to be used as data collection tools in the study.

The women included in the study sample will be divided into two groups as experimental and control groups according to randomization. Experimental group; the group to be trained. control group; This is the group in which no attempt will be made other than data collection.

Statistical Analysis of Data: The data obtained in the research will be analyzed using SPSS (Statistical Package for Social Sciences) for Windows 25.0 program. Homogeneity of descriptive features between groups will be tested by chi-square analysis and independent group t-test. The differentiation status of the scales between the groups will be analyzed with the independent group t-test and the changes within the group will be analyzed with the repeated measures ANOVA test.

ELIGIBILITY:
Inclusion Criteria:

* Be over 18 years old
* Able to speak, read and understand Turkish
* Being scheduled for surgery due to a diagnosis of gynecological cancer
* Having internet access
* Using a smartphone

Exclusion Criteria:

- Having a diagnosis of active psychiatric illness

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
The education given with the mobile application in gynecological oncology patients positively affects the quality of life of the patients. | Women will be evaluated two weeks after surgery.
  The patients' quality of life will be measured with Functional Assessment of Cancer Therapy-General (FACT-G). All questions are aimed at assessing the patients' quality of life in the last 7 days. A higher score from the scale indicates a better quality of life.

SECONDARY OUTCOMES:
Education given with mobile application in gynecological oncology patients positively affects symptom control of patients. | Women will be evaluated two weeks after surgery.
  The patients' symptom will be measured with Symptom Evaluation Form. The symptom evaluation form was created by the researchers by scanning the relevant literature and determining the most common postoperative symptoms of patients who underwent gynecological oncology surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Çisem Baştarcan, Principal Investigator — PhD student
Locations (1):
- Istanbul University-Cerrahpasa, Avcılar, Istanbul, Turkey (Türkiye)